CLINICAL TRIAL: NCT07383636
Title: Comparison of the Plaque Removal Efficacy of Manual and Powered Toothbrushes in Patients Undergoing Clear Aligner Therapy
Brief Title: Comparison of Plaque Removal Efficacy of Different Toothbrushes in Clear Aligner Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Kübra Arslan Çarpar, Assistant Professor, Department of Orthodontics, Faculty of Dentistry, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/1110
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Dental Plaque Accumulation; Oral Hygiene in Orthodontic Patients; Clear Aligner Therapy
Keywords: Clear aligner; Orthodontic attachments; Dental plaque; Plaque index; Oral hygiene; Manual toothbrush; Powered toothbrush; Plaque removal; Orthodontic patients
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: a manual toothbrush group or an electronic toothbrush group. Each participant received only the allocated intervention, and plaque scores were evaluated before and after a single supervised brushing session.
Masking Description: This is an open-label study; no participants, investigators, care providers, or outcome assessors were masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Toothbrush Group (Experimental): Participants brushed their teeth for 2 minutes using a manual toothbrush following standardized oral hygiene instructions during a routine orthodontic visit.
  Interventions: Device: Manual Toothbrush
- Powered Toothbrush Group (Experimental): Participants brushed their teeth for 2 minutes using a powered toothbrush following standardized oral hygiene instructions during a routine orthodontic visit.
  Interventions: Device: Powered Toothbrush

INTERVENTIONS:
Device: Manual Toothbrush — Use of a manual toothbrush for plaque removal in patients undergoing clear aligner therapy.
  Other Names: TePe Select™ Medium
  Arms: Manual Toothbrush Group
Device: Powered Toothbrush — Use of a powered toothbrush for plaque removal in patients undergoing clear aligner therapy.
  Other Names: Oral-B iO 9; Electric toothbrush
  Arms: Powered Toothbrush Group

SUMMARY:
This study aims to compare the effectiveness of manual and powered toothbrushes in removing dental plaque in patients undergoing clear aligner orthodontic treatment.

Clear aligner treatment uses attachments bonded to teeth to facilitate tooth movement. These attachments may increase plaque accumulation around the tooth surface. Poor plaque control can lead to dental caries and periodontal problems.

In this study, patients receiving clear aligner treatment will brush their teeth using either a manual or a powered toothbrush. Dental plaque levels around attachments will be evaluated before and after brushing using a modified plaque index.

The results of this study may help determine whether one type of toothbrush is more effective than the other in maintaining oral hygiene during clear aligner therapy.

DETAILED DESCRIPTION:
Dental plaque is a complex biofilm and a primary etiological factor in the development of dental caries and periodontal diseases. Orthodontic treatments may increase plaque accumulation due to the presence of attachments bonded to the tooth surface.

Clear aligner therapy has become increasingly popular due to its esthetic and removable nature. However, attachments used during treatment may compromise oral hygiene by promoting plaque retention, particularly in the gingival region.

This study is designed to evaluate and compare the plaque removal effectiveness of manual and powered toothbrushes in patients undergoing clear aligner orthodontic treatment.

A total of 14 patients receiving clear aligner therapy will be randomly assigned to either a manual toothbrush group or a powered toothbrush group. Dental plaque accumulation around attachments will be assessed before brushing (T0) and after a standardized two-minute brushing period (T1) using the Modified Plaque Index adapted for orthodontic patients.

Plaque scores will be evaluated at multiple tooth surfaces (mesial, distal, occlusal, and gingival) and analyzed both on a patient-based and tooth-based level. Attachments will also be categorized as conventional or optimized, and plaque reduction will be compared between attachment types.

The findings of this study are expected to provide evidence regarding the effectiveness of different toothbrush types in maintaining oral hygiene in patients treated with clear aligners.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing orthodontic treatment with clear aligners
* Presence of bonded attachments on teeth
* No known systemic diseases
* Not using any regular systemic medications
* Right-handed individuals (actively using the right hand)

Exclusion Criteria:

* Age < 18 years
* Absence of attachments on teeth
* Presence of any systemic disease
* Regular use of systemic medications
* Left-handed or ambidextrous individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2025-11-03 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Modified Plaque Index (MPI) Score After Toothbrushing | Immediately before and immediately after a single 2-minute toothbrushing session
  The primary outcome is the change in dental plaque accumulation measured using the Modified Plaque Index (MPI). Plaque scores will be recorded immediately before toothbrushing (T0) and immediately after a standardized 2-minute toothbrushing session (T1). The difference between T0 and T1 MPI scores will be calculated to assess plaque removal effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Arslan Çarpar, DDS, PhD, Principal Investigator — Mersin University, Faculty of Dentistry, Department of Orthodontics
Locations (1):
- Mersin University, Faculty of Dentistry, Department of Orthodontics, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the small sample size of the study and the potential risk of participant re-identification. Additionally, the informed consent obtained from participants did not include provisions for data sharing beyond the scope of the present study.